CLINICAL TRIAL: NCT04961619
Title: A Real-life Study to Evaluate the Use of Adjuvant Treatment With Dabrafenib and Trametinib in Routine Practice in Patients With Completely Resected High-risk Stage III Melanoma
Brief Title: Adjuvant Dabrafenib and Trametinib Treatment in Patients With Completely Resected High-risk Stage III Melanoma.
Acronym: LEAD Melanoma
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CDRB436BTR01
Record Dates: First submitted 2021-07-05; First posted 2021-07-14 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Melanoma
Keywords: Melanoma; stage III melanoma; BRAF V600E mutation; dabrafenib; trametinib; Turkey
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dabrafenib and trametinib: patients on adjuvant treatment with dabrafenib + trametinib
  Interventions: Drug: dabrafenib; Drug: trametinib

INTERVENTIONS:
Drug: dabrafenib — There was no treatment allocation. Patients administered dabrafenib by prescription that started before inclusion of the patient into the study were enrolled.
Drug: trametinib — There was no treatment allocation. Patients administered trametinib by prescription that started before inclusion of the patient into the study were enrolled.

SUMMARY:
Non-interventional (observational) cohort prospective real life study with primary and secondary data collection from patients on adjuvant treatment with dabrafenib + trametinib in patients with completely resected high-risk stage III (stage IIIA [lymph node > 1mm], IIIB, IIIC and IIID according to AJCC 8th edition) melanoma in Turkey.

DETAILED DESCRIPTION:
The prospective registration of completely resected high-risk stage III melanoma patients treated with dabrafenib and trametinib in the adjuvant setting was based on collaboration with centers of excellence on melanoma patients treatment. Pre-identified centers considered as the most advanced according to their knowledge and experience, took part in the patients recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete surgical resection of histologically confirmed AJCC (8th edition) clinical stage III (stage IIIA [lymph node > 1mm],, IIIB, IIIC, IIID) melanoma, in whom a decision for adjuvant treatment with dabrafenib and trametinib has been made before entering the study;
* V600E mutation-positive cutaneous melanoma;
* ≥ 18 years of age;
* Written informed consent signed.

Exclusion Criteria:

* Lack of basic demographic and staging data.
* Current active participation in an interventional clinical trial for treatment of melanoma.
* Pregnancy or breastfeeding women.
* Current primary diagnosis of a cancer other than melanoma, that requires systemic or other treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Completely resected high-risk stage III melanoma patients treated with dabrafenib and trametinib in the adjuvant setting
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Relapse-free survival (RFS) rate | 12 months
  RFS is the length of time after primary treatment for a cancer ends that the patient survives without any signs or symptoms of that cancer.

SECONDARY OUTCOMES:
Total duration of treatment | until end of treatment or permanent treatment discontinuation
  Total duration of treatment defined as median time on adjuvant dabrafenib + trametinib treatment (from start to end of treatment/permanent treatment discontinuation).
Number of patients on treatment | Baseline, up to 12 months
  Collection of number of patients on treatment
Rate of permanent study drug discontinuation | 12 months
  Rate of permanent study drug discontinuation due to any reason
Rate of permanent drug discontinuation due to pyrexia and other AEs | 12 months
  Rate of permanent drug discontinuation due to pyrexia and other AEs
incidence and severity of Adverse Events (AEs) | 12 months
  Collection of incidence and severity of Adverse Events
procedures of the management of Adverse Events (AEs) | 12 months
  Collection of procedures of the management of Adverse Events (AEs)
Reason for treatment discontinuation | 12 months
  death, relapse, AEs, withdrawal of consent, other
Average dose of dabrafenib and trametinib used during the treatment | 12 months
  Average dose of dabrafenib and trametinib used during the treatment including dose reductions.
Proportion of patients with dabrafenib and trametinib dose reduction during treatment | 12 months
  collection of the proportion of patients with dabrafenib and trametinib dose reduction during treatment
Reason for dabrafenib and trametinib dose reduction | 12 months
  Collection of the reason for dabrafenib and trametinib dose reduction
Time since surgery | 12 months
  Collection of the time since surgery
Type of relapse | 12 months
  Collection of the type of relapse: local, regional or distant

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Turkey (Türkiye) (9):
  - Novartis Investigative Site, Antalya, Konyaalti
  - Novartis Investigative Site, Edirne, Merkez
  - Novartis Investigative Site, Bursa, Nilufer
  - Novartis Investigative Site, Diyarbakır, Sur
  - Novartis Investigative Site, Istanbul, Uskudar
  - Novartis Investigative Site, Adana, Yuregir
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Kecioren Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18387